CLINICAL TRIAL: NCT02363972
Title: Ellipsys Vascular Access Catheter System Clinical Trial
Brief Title: Percutaneous Less Invasive AV Fistula for Vascular Access in ESRD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-0014-01
Record Dates: First submitted 2015-02-06; First posted 2015-02-16 (Estimated); Results first posted 2020-09-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: End Stage Renal Disease; AV Fistula; Fistula; End Stage Kidney Disease
MeSH Terms: conditions — Kidney Failure, Chronic; Arteriovenous Fistula; Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ellipsys Vascular Access Catheter (Experimental): ESRD patients who require and qualify for creation of a surgical AV fistula will be offered the opportunity to participate in this study for a less invasive way of creating an AV fistula.
  Interventions: Device: Ellipsys Vascular Access Catheter

INTERVENTIONS:
Device: Ellipsys Vascular Access Catheter — A one-time use vascular catheter used as a less invasive means of creating an AV fistula. Screening and follow-up assessments are standard of care for surgical AV fistulae.

SUMMARY:
A prospective single-arm well-controlled study to evaluate the safety and effectiveness of a less invasive means of establishing vascular access to facilitate dialysis in patients with end stage renal disease.

ELIGIBILITY:
Inclusion Criteria:

Patients were eligible for enrollment into the study if they met the following criteria:

1. Patients ≥ 18 years of age and ≤ 80 years of age
2. Male or non-pregnant female (verified with a urine/blood pregnancy test, for women of reproductive potential)
3. Life expectancy of at least one year, per the investigator's opinion
4. Diagnosed with end-stage renal disease (ESRD) or chronic kidney disease requiring dialysis or anticipated start of dialysis within 6 months of enrollment
5. Patients deemed medically eligible for upper extremity autogenous AV fistula creation, per institutional guidelines and/or clinical judgment
6. Adequate quality vein based on pre-operative assessment

   1. Adjacent vein diameter of ≥ 2.0 mm at target anastomosis site
   2. Confirmed clinically significant outflow
7. Adequate quality radial artery based on pre-operative assessment

   a. Arterial lumen diameter of ≥ 2.0 mm at target anastomosis site
8. Adequate collateral arterial perfusion

   1. Patent palmar arch
   2. Negative Allen's Test for ulnar artery insufficiency
9. No clinical evidence of subclavian artery stenosis on the ipsilateral side.
10. Radial artery-adjacent vein proximity ≤ 1.5 mm measured lumen edge-to-lumen edge as determined by pre-procedural ultrasound and confirmed pre-procedure
11. Patient was able to provide written informed consent
12. Able to travel to enrolling institution for follow-up examinations
13. Able and willing to follow a daily aspirin and/or other anti-coagulation/antiplatelet regimen, not including warfarin (Coumadin, or comparable anti-coagulant, see exclusion criteria 15)

Exclusion Criteria:

Patients were excluded if any of the following was true:

1. Documented or suspected central venous stenosis including upper extremity arterial stenosis (≥ 50%)
2. a. Prior vascular surgery at or proximal (central) to the AVF target site b. Prior axillary dissection or mastectomy on the ipsilateral side as intended AV fistula site
3. History of steal syndrome from a previous hemodialysis vascular access on the ipsilateral side which required intervention or abandonment
4. Evidence of vascular disease at the radial artery/adjacent vein site on the ipsilateral side
5. Pre-existing vascular disease that could confound the study results
6. Systolic pressures < 100 mm Hg at the time of screening
7. Suspected or confirmed skin disease at the skin entry site
8. Immunocompromised patients (e.g. HIV positive)
9. Edema of the upper extremity on the ipsilateral side
10. Patients requiring immunosuppressant therapy such as sirolimus (Rapamune®) or Prednisone at a dose of > 10 mg per day
11. Peripheral white blood cell count < 1.5 K/mm3 or platelet count < 75,000 cells/mm3
12. Current diagnosis of carcinoma (defined as in remission < 1 year)
13. Pregnant or currently breast feeding
14. Known bleeding diathesis or coagulation disorder
15. Receiving warfarin (Coumadin, or comparable anti-coagulant) therapy
16. Patients with acute or active infection
17. Scheduled kidney transplant within 6 months of enrollment
18. Participation in another clinical investigation (excluding retrospective studies or studies not requiring a consent form)
19. History of substance abuse or anticipated to be non-compliant with medical care or study requirements based on investigator judgment
20. Patient required creation of an arteriovenous fistula distal to the wrist
21. Patient required nerve block requiring immobilization of the arm

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2015-02-10 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Hull, MD, Principal Investigator — Richmond Vascular Center
Locations (5):
- United States (5):
  - Southwest Vascular Center, Tempe, Arizona
  - BNMG San Diego Vascular Access Center, San Diego, California
  - Dallas Nephrology Associates, Plano, Texas
  - San Antonio Kidney Disease Center, San Antonio, Texas
  - Richmond Vascular Center, North Chesterfield, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ellipsys Vascular Access Catheter
Started | 103
Completed | 77
Not Completed | 26

BASELINE CHARACTERISTICS:
Arm/Group | Ellipsys Vascular Access Catheter
Number analyzed (Participants) | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37
  Not Hispanic or Latino | 65
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 21
  White | 77
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Maturation Success Rate at 90 Days
Description: Maturation success rate of the access site was a binary endpoint defined as (1) achievement of a venous diameter of greater than or equal to 4 mm and (2) blood flow greater than or equal to 500 ml/min as measured via duplex ultrasound at the 90 day follow-up visit for the ITT population.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ellipsys Vascular Access Catheter
Number analyzed (Participants) | 103
Participants | 92

2. Primary Outcome: Number of Participants With Device-related Serious Adverse Events
Description: The primary safety endpoint was defined as the percent of subjects having one or more of the following device-related serious adverse events: vessel perforation, vessel dissection, and electrical shock during index; and significant embolization in a previously uninvolved arterial territory within 90 days of the index procedure.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ellipsys Vascular Access Catheter
Number analyzed (Participants) | 103
Participants | 0

3. Secondary Outcome: Percent of Participants With Access Systems That Successfully Created an AVF
Description: Percent of Ellipsys Vascular Access Systems that successfully created an AVF upon deployment
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ellipsys Vascular Access Catheter
Number analyzed (Participants) | 103
Participants | 102

4. Secondary Outcome: Percent of Access Sites With Clinical Patency at Discharge
Description: Percent of access sites that demonstrated physical exam patency through clinic discharge
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ellipsys Vascular Access Catheter
Number analyzed (Participants) | 102
Participants | 98

5. Secondary Outcome: Percent of Access Sites That Sustain 2-needle Cannulation by 90 Days
Description: Percent of access sites that could sustain three 2-needle cannulations at the prescribed needle gauge and blood flow rate (Qb) between the 4 week and 90 day follow-up visits after initial AV fistula creation
Time Frame: 90 days
Population: The analysis population analyzed (65) is a subset of of the overall number of participants analyzed (103) due to not all participants being on dialysis an requiring 2 needle cannulation by the 90 day outcome measure time frame
Measure: Count of Participants; unit: Participants
Arm/Group | Ellipsys Vascular Access Catheter
Number analyzed (Participants) | 65
Participants | 29

6. Secondary Outcome: Percent of Access Sites That Achieved or Maintained Maturation at 90 Days
Description: Percent of access sites which achieved or maintained maturation following intervening manipulations (surgical or endovascular) designed to promote or reestablish maturation. This definition also includes common definition for secondary patency.
Time Frame: 90 days
Population: The analysis population analyzed (102) is a subset of of the overall number of participants analyzed (103) due to not all participants having a patent fistula at discharge from the index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Ellipsys Vascular Access Catheter
Number analyzed (Participants) | 102
Participants | 85

7. Secondary Outcome: Percent of Access Sites That Achieved Maturation Without Intervention
Description: Percent of access sites that achieved and maintained maturation without any surgical or endovascular intervention designed to promote or reestablish maturation
Time Frame: 90 days
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Ellipsys Vascular Access Catheter
Number analyzed (Participants) | 102
Participants | 1

8. Secondary Outcome: Percent of Access Sites That Were Patent Following Intervention
Description: Percent of access sites which were patent after intervening manipulations (surgical or endovascular) intended to promote or reestablish patency
Time Frame: 90 days
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Ellipsys Vascular Access Catheter
Number analyzed (Participants) | 102
Participants | 89

9. Secondary Outcome: Percent of Access Sites That Achieved Patency Without Intervention
Description: Percent of access sites that maintained patency without any surgical or endovascular intervention designed to maintain or reestablish blood flow in the access site
Time Frame: 90 days
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Ellipsys Vascular Access Catheter
Number analyzed (Participants) | 102
Participants | 1

10. Secondary Outcome: Intervention Rate
Description: Percent of subjects who had one or more surgical or endovascular interventions to maintain or reestablish blood flow in the access site
Time Frame: 90 days
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Ellipsys Vascular Access Catheter
Number analyzed (Participants) | 102
Participants | 98

11. Secondary Outcome: Transposition Rate
Description: Percent of subjects who required one or more surgical transpositions performed to facilitate needle access
Time Frame: 90 days
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Ellipsys Vascular Access Catheter
Number analyzed (Participants) | 102
Participants | 19

12. Other Pre Specified Outcome: Time to First AVF Cannulation
Description: Time to AVF cannulation was defined as the elapsed time to the first use of access site (from the date of the study procedure).
Time Frame: 90 days
Population: The analysis population analyzed (33) is a subset of of the overall number of participants analyzed (103) due to not all participants having a patent fistula at discharge from the index procedure and not requiring cannulation by the 90 day outcome timeframe
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Ellipsys Vascular Access Catheter
Number analyzed (Participants) | 33
Days | 67.8 (15.9)

13. Other Pre Specified Outcome: Catheter Utilization
Description: Catheter utilization was defined as the total number of days a catheter was used before access site maturation per subject. The start date was either 1) the date of the study procedure, for subjects who already had a dialysis catheter in place or 2) the date placed, if during the study. The end date was either 1) the date the catheter was removed or 2) the 90 day visit, if the catheter was still in place.
Time Frame: 90 days
Population: The analysis population analyzed (32) is a subset of of the overall number of participants analyzed (103) due to not all participants having a patent fistula at discharge from the index procedure and not requiring a catheter utilization by the 90 day outcome timeframe
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Ellipsys Vascular Access Catheter
Number analyzed (Participants) | 32
days | 83.1 (17.4)

14. Other Pre Specified Outcome: Target Vessel Location
Description: Anatomic location of matured target vessel
Time Frame: 90 days
Population: The analysis population analyzed (90) is a subset of of the overall number of participants analyzed (103) due to not all participants having a patent fistula at discharge from the index procedure and not achieving an identifiable target vein by the 90 day outcome timeframe
Measure: Count of Participants; unit: Participants
Arm/Group | Ellipsys Vascular Access Catheter
Number analyzed (Participants) | 90
Participants
  Cephalic vein | 68
  Basilic vein | 20
  Brachial vein 1 | 1
  Brachial vein 2 | 1

ADVERSE EVENTS:
Time Frame: 90 days
Description: Serious Adverse Events and Other Adverse Events were monitored/assessed without regard to the specific Adverse Event Term.
Arm/Group | Ellipsys Vascular Access Catheter
Serious Adverse Events (participants affected / at risk) | 18/103
Other Adverse Events (participants affected / at risk) | 28/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ellipsys Vascular Access Catheter (N=103)
Cardiac serious adverse events (Cardiac disorders) | 4
Endocrine, metabolic nutritional serious adverse events (Endocrine disorders) | 1
Gastrointestinal serious adverse events (Gastrointestinal disorders) | 2
Musculoskeletal serious adverse events (Musculoskeletal and connective tissue disorders) | 2
Nervous system serious adverse events (Nervous system disorders) | 1
Respiratory serious adverse events (Respiratory, thoracic and mediastinal disorders) | 2
Skin and subcutaneous serious adverse events (Skin and subcutaneous tissue disorders) | 1
Vascular, blood and lymphatic serious adverse events (Vascular disorders) | 4
Uncoded (Social circumstances) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ellipsys Vascular Access Catheter (N=103)
Eye, ear nonserious events (Ear and labyrinth disorders) | 1
Immune, infection nonserious events (Immune system disorders) | 3
musculoskeletal nonserious adverse events (Musculoskeletal and connective tissue disorders) | 3
Skin nonserious adverse events (Skin and subcutaneous tissue disorders) | 2
Surgical procedure nonserious adverse events (Surgical and medical procedures) | 1
Vascular, blood nonserious adverse events (Vascular disorders) | 17
Drug effect nonserious adverse events (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No